CLINICAL TRIAL: NCT07138664
Title: Promoting Mental Health Among At-risk Adolescents in Malaysia
Acronym: MyHeRo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Collaborators: Universiti Malaysia Sabah (Other); University Malaysia Sarawak (Other); Universidad Complutense de Madrid (Other); Sunway University (Other); Saglik Bilimleri Universitesi (Other); University of Exeter (Other); University of Malaya (Other); National University of Malaysia (Other)
Responsible Party: Principal Investigator, Cecilia Essau, Professor of Developmental Psychopathology, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSYC 23-483
Record Dates: First submitted 2025-08-16; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Depression in Adolescence; Anxiety
Keywords: Anxiety; Depression; Adolescents; School-based intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Super Skills for Life program (Experimental): A manualized psychosocial program for preventing anxiety and depression and for promoting healthy lifestyles (called "Super Skills for Life; SSL"). SSL focuses on: (1) teaching about healthy lifestyles; (2) building emotional resilience through stress management; (3) encouraging peer learning and building peer networks; and (4) promoting self-confidence and social skills. These key elements are organized over 8 weekly sessions in a group format (45-60 minutes per session).
  Interventions: Behavioral: Super Skills for Life program
- Study-Skills program (Experimental): Study-Skills program will be implemented in a group format (45-60 minutes per session) in 8 weekly sessions, covering: note-taking skills, effective study strategies, and time management.
  Interventions: Behavioral: Study-Skills program

INTERVENTIONS:
Behavioral: Super Skills for Life program — Study-Skills program will be implemented in a group format (45-60 minutes per session) in 8 weekly sessions, covering: note-taking skills, effective study strategies, and time management.
  Other Names: Study-Skills program
  Arms: Super Skills for Life program
Behavioral: Study-Skills program — Study-Skills program will be used as a comparator intervention, which will be implemented in a group format (45-60 minutes per session) in 8 weekly sessions, covering: note-taking skills, effective study strategies, and time management.
  Arms: Study-Skills program

SUMMARY:
The primary objective of this trial is to evaluate a school-based intervention designed to promote mental health among at-risk adolescents from low-income communities in Malaysia. The study will employ a two-arm, cluster randomised controlled trial design, comparing a school-based intervention to a control condition. Adolescents will be recruited from at least 20 secondary schools located in economically disadvantaged rural and urban areas of Malaysia. Assessments will take place at multiple time points: during screening, at baseline (pre-intervention), immediately after the intervention (8 weeks), and at two follow-up points-6 and 12 months post-intervention. The primary outcomes are a reduction in anxiety and depressive symptoms, along with improved mental wellbeing at the 12-month follow-up.

DETAILED DESCRIPTION:
The overall aim of this trial is to use a school-based intervention to promote mental health among at-risk adolescents from low-income communities in Malaysia. Our primary aim is to evaluate the effectiveness and cost-effectiveness of a school-based intervention ("Super Skills for Life"; SSL) in reducing anxiety and depression, and in improving mental wellbeing in adolescents aged 12-14 years. We also aim to identify contextual factors related to the successful implementation of SSL in Malaysian schools.

This study will use a two-arm, cluster randomised controlled trial design with a 1:1 allocation ratio to compare a school-based intervention (Super Skills for Life; SSL) to a control condition (Study Skills Programme; SSP). Three stratification factors will be used for randomisation: school size, classes/forms and school location (urban vs rural). These adolescents will be invited to complete a screening questionnaire (i.e., Depression Anxiety and Stress Scale-21; DASS-21).

Based on power calculations, a total of 428 adolescents (214 per arm) with moderate to severe symptoms of anxiety and depression will be recruited to participate in the trial. Classrooms will be randomly assigned to either the intervention or control group, and eligible adolescents within each class will receive the intervention assigned to their group. Assessments will be conducted at screening, baseline (pre-intervention), immediately after the intervention (8 weeks), and at two follow-up points-6 and 12 months post-intervention. The primary outcomes will include reductions in anxiety and depressive symptoms, along with improvements in mental wellbeing at the 12-month follow-up.

Findings of this trial will determine if delivering a group school-based intervention by school staff for adolescents at risk of anxiety and depression is effective and cost-effective.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent (aged 12-14) who are in the first two years (Form 1 and Form 2, equivalent to year 7 and 8 in the United Kingdom school system, respectively) in lower secondary schools.
2. Adolescents score moderate to severe levels of anxiety and/or depression on the Depression Anxiety and Stress Scale-21 (DASS-21) based on the original cut-off norms (DASS-21 Anxiety scale ≥ 10 and/or DASS-21 Depression scale ≥ 14).
3. Adolescent's parent/carer provides written consent.

Exclusion Criteria:

(1) Being diagnosed with neurodevelopmental disorders. (2) Being diagnosed with intellectual disability.

-

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 428 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in adolescent's anxiety and depression | Pre-intervention, as well as at 8 weeks, and at 6 and 12 months after the intervention.
  The Revised Children's Anxiety and Depression Scale will be used to identify symptoms of anxiety and depressive disorder in adolescents. It contains 6 items for measuring anxiety and 5 items for depression symptoms, which are to be rated on a 4-point Likert Scale from 0 ("never") to 3 ("always").
Change in adolescent's wellbeing | Pre-intervention, as well as at 8 weeks, and at 6 and 12 months after the intervention.
  Short Warwick-Edinburgh Mental Well-being Scale will be used to measure mental wellbeing. All its 7 items are worded positively and cover feeling and functioning aspects of mental wellbeing. The items can be rated on a 5-point scale from 1 (none of the time) to 5 (all of the time).

SECONDARY OUTCOMES:
Change in adolescent's emotion regulation strategies. | Pre-intervention, as well as at 8 weeks, and at 12 months after the intervention.
  Cognitive Emotion Regulation Questionnaire will be used to measure emotion regulation strategies. It consists of 18 items, which can be rated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always) in response to how often each of the 9 emotion regulation strategies are used: refocus on planning, putting into perspective, acceptance, positive refocusing, positive reappraisal, self-blame, other blame, rumination, and catastrophizing.
Change in adolescent's suicidal behaviour. | Pre-intervention, as well as at 8 weeks, and at 12 months after the intervention.
  The Paykel Suicide Scale (PSS) will be used to measure suicidal behaviour. The scale consists of 5 items, with a dichotomous response system, i.e., Yes or No.
Change in adolescent's ability to carry out essential social behaviors. | Pre-intervention, as well as at 8 weeks, and at 6 and 12 months after the intervention.
  The Social Skills Questionnaire will be used to measure essential social behaviors that contribute to success in social interactions. Its 13 items can be are rated from 0 (Not true), 1 (Sometimes true) to 2 (Mostly true).
Change in adolescent's working memory and inhibition. | Pre-intervention, as well as at 8 weeks, and at 12 months after the intervention.
  Teenage Executive Functioning Inventory will be used to measure working memory and inhibition. It contains 20 items which can be rated on a 5-point Likert scale ranging from 1 ("definitely not true") to 5 ("definitely true").
Change in adolescent's executive function. | Pre-intervention, as well as at 8 weeks, and at 12 months after the intervention.
  Executive function will also be measured using milliseconds experimental task to measure attention control and working memory.
Change in the severity of anxiety and depressive symptoms. | Pre-intervention, as well as at 8 weeks, and at 12 months after the intervention.
  Depression Anxiety and Stress Scale-21 (DASS-21) will be used to measure adolescent's severity of anxiety and depressive symptoms. The DASS-21 consists of 21 items which are divided equally across the anxiety, depressive and stress subscales, which can be rated on a 4-point Likert Scale (range from 0 [did not apply to me at all] to 3 [applied to me very much or most of the time]).
Change in adolescent's lifestyle habits. | Pre-intervention, as well as at 8 weeks, and at 6 and 12 months after the intervention.
  Lifestyle and Habits Questionnaire (LHQ-B) will be used to measure adolescent's lifestyle habits (physical activity and exercise, sleep and sleep hygiene, and type of food consumption).
  LHQ-B contains 16 items which ask adolescents about how frequently they perform each behaviour in the past 30 days on a 5-point scale from "never" to "always".

OTHER OUTCOMES:
Changes in adolescent's self-esteem. | Pre-intervention, as well as at 8 weeks, and at 12 months after the intervention.
  Rosenberg Self-Esteem Scale (RSES) will be used to measure global self-worth. Three out of 10 items will be used in the present study, which can be rated on a 4-point Likert scale format ranging from 4 (strongly agree) to 1 (strongly disagree).
Changes in adolescent's academic stress. | Pre-intervention, as well as at 8 weeks, and at 6 and 12 months after the intervention.
  The Educational Stress Scale for Adolescents will be used to measure adolescent's perceived academic stress. Its 16 statements can be rated on a five-point Likert scale ranging from "strongly disagree" to "strongly agree".
Changes in adolescents' feelings about their school and teachers. | Pre-intervention, as well as at 8 weeks, and at 12 months after the intervention.
  School Connectedness Scale will be used to adolescents' feelings about their school and teachers. Its 5 items can be rated on a five-point response format ranging from 0 (Strongly disagree) to 4 (Strongly agree).
Measure facilitators' attitudes toward the adoption of evidence-based practices. | Pre-intervention.
  Evidence-based Practice Attitude Scale for Teachers will be used to measure facilitators' attitudes toward the adoption of evidence-based practices (EBPs). It contains 13 items can be rated on a 5-Likert scale, ranging from "Not at All" (0) to "To a Very Great Extent" (4).
Changes in adolescent's health-related quality of life. | Pre-intervention and at 12 months after the intervention.
  The Child Health Utility will be used to measure health-related quality of life. It consists of 9 domains (worry, sadness, pain, tiredness, annoyance, school, sleep, daily routine and activities), and within each dimension, there are five different levels with increasing levels of severity.
Changes in parent's quality of life, cost-utility of healthcare interventions, and computation of quality-adjusted life years. | Pre-intervention and at 12 months after the intervention.
  Self-reported European Quality of Life Five Dimension will be used to measure parent's quality of life, cost-utility of healthcare interventions, and computation of quality-adjusted life years.
Changes in cost incurred by adolescents across healthcare, social care and community settings. | Pre-intervention and at 12 months after the intervention.
  Client Service Receipt Inventory to collect information from the parents related to cost-related data, by estimating associated costs across healthcare, social care and community settings. Parent will further be asked about adolescent's frequency and cost of using mental and physical health and social services.

CONTACTS AND LOCATIONS:
Locations (5):
- Malaysia (5):
  - Fakulti Psikologi Dan Pendidikan, Kota Kinabalu, Sabah
  - Universiti Malaysia Sarawak, Kuching, Sarawak
  - Universiti Kebangsaan Malaysia, Bangi, Selangor
  - Universiti Malaya, Kuala Lumpur, Selangor
  - Sunway University, Subang Jaya, Selangor

IPD SHARING:
Plan to Share IPD: No
Data will not be shared on an individual basis. Anonymised study data will be archived at the end of the study through the University of Roehampton data repository.

REFERENCES:
- [Derived] Essau CA, Zakaria S, Ting CH, Lee JAC, de la Torre-Luque A, Ng ALO, Majid HA, Dodd H, Nik Farid ND, Muhammad NA, Wahab S. Promoting mental health among at-risk adolescents in Malaysia (MyHeRo): study protocol for a cluster randomised controlled trial to evaluate the effectiveness and cost-effectiveness of a school-based intervention compared with study skills condition for adolescents identified as at risk for anxiety and depression. Trials. 2026 Jan 28. doi: 10.1186/s13063-025-09368-7. Online ahead of print. PMID 41593785